CLINICAL TRIAL: NCT05705245
Title: The Effect of Alveolar Recruitment Maneuver on Perioperative Oxygenation, Oxygen Reserve Index (ORi) and Postoperative Pulmonary Complications in Morbid Obese Patients Undergoing Laparoscopic Bariatric Surgery
Brief Title: Effects of Recruitment Manouever on Oxygenation, Oxygen Reserve Index and Postoperative Pulmonary Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, hafize fisun demir, assistant professor, Balikesir University
Other Study IDs: 2021/138
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: obesity, bariatric surgery, alveolar recruitment, oxygen reserve index
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recruitment: Patients who received alveolar recruitment manouever during bariatric surgery
  Interventions: Other: recruitment
- non recruitment: patients who did not receive alveolar recruitment manoeuver during bariatric surgery

INTERVENTIONS:
Other: recruitment — Automated alveolar recruitment menouever applied during mechanical ventilation in the intraoperative period
  Groups: recruitment

SUMMARY:
General anesthesia and mechanical ventilation decrease pulmonar volume; attenuate small airway closure, atelectasis, and increase the rate of hypoxia and postoperative pulmonary complications. Lung volume in obese patients decreases inversely with the increase in body mass index. Obesity is associated with increased atelectasis, hypoxia and postoperative pulmonary complication rates during anesthesia . Alveolar recruitment maneuver is a technique where high positive end-expiratory pressure (PEEP) is applied for for short periods, follwed by a continuous PEEP appşication throughout surgery. This has become a standard practice during anesthesia in recent years. Oxygen reserve index (ORi) is an index measured with a non-invasive finger-tip sensor and shows the oxygen content of the venous blood. It is effective at high oxygen levels and may indicate the presence of hyperoxia. Our aim is to examine the effect of alveolar recruitment maneuver on oxygenation parameters under anesthesia and the correlation with ORi in morbidly obese patients.

DETAILED DESCRIPTION:
Patients with body mass index> 40 m2, scheduled for bariatric surgery under general anesthesia will be monitorised with the ORi sensor and monitored at regular intervals. Preoperative and postoperative lung aeration will be evaluated with lung ultrasaund. İntraoperative standart anesthesia will be administered by an anesthesiolıgist not aware of the ultrasound. Alveolar recruitment will be applied by the same anesthesiologist if necessary. Blood gas samples obtained throughout surgery will be evaluated. ORİ values and intraoperative vital, respiratory, neuromuscular monitoring parameters will be obtained. Postoperative pulmonary complicationsa will be evaluated at postoperative day 5.

Finding will be compared between patients who received recruitment and who did not.

ELIGIBILITY:
Inclusion Criteria:

Bariatric surgery general anesthesia and mechanical ventilation via orotracheal entubation Age between 18-65 ASA I-III BMI > 40 m-2

Exclusion Criteria:

Previous history of thorasic surgery, pneumothorax Chemo or Radiotherapy to the chest within 2 months History of Respiratory disease (COPD, emphysema, pneumonia, lung malignancy, Lung Bulla ) Emergency surgery Cardiovascular, renal, hepatic, neuromuscular disease İntracrabial pathology or trauma High intraoptic pressure Pulmonary Hypertension Pregnancy Criticall illness, or history of mechanical ventilation within 1 month

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: obese patients with BMI> 40 scheduşed for bariatric surgery
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complications | 5 days
  Coughing, dyspnoe, side pain, phlegm

SECONDARY OUTCOMES:
Effect of recruitment manoeuver on oxygene reserve index | intraoperative
  oxygene reserve index measured through a digital probe

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University Hospital, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no plan to sharing